CLINICAL TRIAL: NCT00538785
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of MEDI-524, a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), in Children With Hemodynamically Significant Congenital Heart Disease
Brief Title: A Study to Evaluate MEDI-524 In Children With Hemodynamically Significant Congenital Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Pamela Griffin, Senior Director, Clinical Development, MedImmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP124-S2; NCT00240890 (obsolete NCT alias)
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Congenital Heart Disease
Keywords: Synagis, motavizumab, palivizumab, children, MEDI-524, RSV, congenital hear disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — motavizumab; Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motavizumab (Experimental): Motavizumab was administered as an intramuscular injection at 15 mg/kg every 30 days during the RSV season for a maximum of 5 scheduled doses. Additionally, children who underwent cardiac surgery with cardiopulmonary bypass through Study Day 150 were to receive a protocol-specified replacement dose of study drug immediately following the surgery when determined by the physician to be medically stable for an IM injection.
  Interventions: Biological: Motavizumab
- Pailvizumab (Active Comparator): Palivizumab was administered as an intramuscular injection at 15 mg/kg every 30 days during the RSV season for a maximum of 5 scheduled doses. Additionally, children who underwent cardiac surgery with cardiopulmonary bypass through Study Day 150 were to receive a protocol-specified replacement dose of study drug immediately following the surgery when determined by the physician to be medically stable for an IM injection.
  Interventions: Biological: Palivizumab

INTERVENTIONS:
Biological: Motavizumab — 15 mg/kg IM administered at monthly intervals
  Other Names: Medi-524
  Arms: Motavizumab
Biological: Palivizumab — 15 mg/kg IM administered at monthly intervals
  Other Names: Synagis
  Arms: Pailvizumab

SUMMARY:
The primary goal was to describe the safety of the investigational product when given monthly to prevent serious respiratory infection among children with significant heart disease.

DETAILED DESCRIPTION:
The primary objective was to describe the safety and tolerability of motavizumab when given monthly as prophylaxis against serious RSV infection among children with hemodynamically significant congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* 24 months of age or younger at randomization (child must have been randomized on or before their 24-month birthday)
* Documented, hemodynamically significant CHD
* Unoperated or partially corrected CHD
* Written informed consent obtained from the patient's parent(s)/legal guardian(s) Note: The following children were not eligible: children with uncomplicated small atrial or ventricular septal defects or patent ductus arteriosus, children with aortic stenosis, pulmonic stenosis, or coarctation of the aorta alone. Children with acyanotic cardiac lesions must have pulmonary hypertension [≥ 40 mmHg measured pressure in the pulmonary artery (PA)] or the need for daily medication to manage CHD.

Exclusion Criteria:

* Unstable cardiac or respiratory status, including cardiac defects so severe that survival was not expected or for which cardiac transplantation was planned or anticipated
* Hospitalization, unless discharge was anticipated within 21 days
* Anticipated cardiac surgery within two weeks of randomization
* Requirement for mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure or other mechanical respiratory or cardiac support
* Associated non-cardiac anomalies or end organ dysfunction resulting in anticipated survival of less than six months or unstable abnormalities of end organ function
* Acute respiratory illness, or other acute infection or illness Note: children with any respiratory symptoms must have had a negative RSV test prior to randomization
* Chronic seizure or evolving or unstable neurologic disorder
* Known immunodeficiency
* Mother with HIV infection (unless the child had been proven to be not infected)
* Known allergy to Ig products
* Receipt of any polyclonal antibody (for example, Hepatitis B IG, IVIG, VZIG) within 3 months prior to randomization
* Receipt of palivizumab (Synagis®) within 3 months prior to randomization
* Use of investigational agents within the past three months (other than investigational agents commonly used during cardiac surgery or the immediate post-operative period, e.g., nitric oxide)
* Current participation in other investigational protocols of drugs or biological agents
* Previous participation in MI-CP124 (Season 1)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1236 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Griffin, 301-398-0000, Study Director — MedImmune LLC
Locations (151):
- United States (30):
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital And Health Center, San Diego, California
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic Biomedical Research Department, Orlando, Florida
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Suny At Stony Brook University Medical Center, Stony Brook, New York
  - Univ. of North Carolina, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Children's Cardiology Associates PLLC, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Austria (3):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Innsbruck
  - Allgemeines Krankenhaus Linz, Linz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Wein
- Belgium (9):
  - Ziekenhuisnetwerk Antwerpen - Koningin Paola Kinderziekenhuis, Antwerp
  - UZ Brussel, Brussells
  - Hôpital Universitaire des Enfants Reine, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
- Bulgaria (8):
  - University Multifunctional Hospital for Active Treatment, Pleven
  - University Mulitiprofile Hospital for Active Treatment "St.Georgi", Plovdiv
  - Multifunctional Hospital for Active Treatment - Pleven, Plovdiv
  - Regional Dispensary for Pulmonary Diseases with Inpatient sector-Rousse, Rousse
  - Specialized Hospital for Active Treatment of Cardio-vascular Diseases, Sofia
  - Specialized Hospital for Active Treatment of Pediatric Diseases, Sofia
  - University Multifunctional Hospital for Active Treatment, Stara Zagora
  - Multifunctional Hospital for Active Treatment - Pleven, Varna
- Canada (8):
  - Children's and Women's Hospital of BC, Room #1R11, Vancouver, British Columbia
  - IWK Health Center, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
  - University of Alberta, Edmonton
  - Montreal Children's Hospital, Montreal
  - Saint Justine Hospital, Montreal
  - Children's Hospital Of Eastern Ontario, Ottawa
  - Saskatchewan Drug Research Institute, Saskatoon SK
- Czechia (7):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Most, prispevkova organizace, Most
  - Fakultni nemocnice Plzen, Plzen - Lochotin
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Ustav pro peci o matku a dite, Prague
  - Fakultni nemocnice v Motole, Prague
  - Fakultni nemocnice Na Bulovce, Prague
- Skejby Sygehus, Århus N, Denmark
- France (8):
  - Groupe Hospitalier Pelligrin, Bordeaux
  - CHRU Dijon-Complex du Bocage, Dijon
  - Centre chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Hospital de la Conception, Marseille
  - Hospital Robert Debre, Paris
  - American Memorial Hospital, Reims
  - Hospital de Hautepierre, Strasbourg
  - Hospitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Friedrich-Alexander-Universiät Erlangen Nürnberg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig Holstein, Kiel
  - Johannes Gutenberg-Universität, Mainz
  - LMU Klinikum der Universität, München
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinik Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (9):
  - Semmelweis Egyetem, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Gyermeksziv Kozpont, Budapest
  - Debreceni Egyetem OEC, Debrecen
  - Petz Aladar Megyei Korhaz, Győr
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Josa Andras Korhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem AOK, Gyermekgyogyaszati Klinika, Szeged
  - Veszprém Megyei Önkormányzat - Csolnoky Ferenc Kórház, Veszprém
- Israel (9):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Lebanon (3):
  - St George University Hospital, Achrafieh- Beirut
  - American University of Beirut Medical Center, Beirut
  - Hotel Dieu De France, Beirut
- Poland (9):
  - Samodzielny Publiczny Szpital Akademii Medycznej, Bialystok
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Wojewodzki Szpital im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Wojewodzki Szpital Dzieciecy W Bydgoszczy, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Dzieciecy Szpital Kliniczny im. Prof. Antoniego Gebal Poliklinika, Lubin
  - Ginekologiczno-Poloznicy Szpital Kliniczny Uniwersytetu Medycznego w Poznaniu, Poznan
  - Szpital Kliniczny Uniwersytetu Medycznego im. Karola Jonschera, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. Tadeusza Sokolowskiego Pomorskiej AM w Szczecinie, Szczecin
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
- Russia (8):
  - Kazan State Medical University, Kazan'
  - Kuban State Medical Academy, Krasnodar
  - Meshalkin Research Institue of Blood circulation, Novosibirsk
  - City Outpatient Clinic #113, Saint Petersburg
  - Saint Petersburg State Pediatric Medical Academy, Saint Petersburg
  - St. Petersburg City Children's Hospital #1, Saint Petersburg
  - Research Cardiology Institute of Tomsk Scientific Center, Tomsk
  - St. Petersburg Pediatric city hospital, Tyumen
- Spain (18):
  - Hospital Juan Canalejo, A Coruña
  - Hospital de Cruces, Barakaldo
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Sant Joan de Deu, Esplugas de Llobregat
  - Hospital Josep Trueta, Girona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Materno Infantil de Jaen, Jaén
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Gregorio Marañon, Madrid
  - Hospital La Paz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Materno Infantil, Málaga
  - Hospital Infantil Universitario Virgen del Rocío, Seville
  - Hospital Xeral de Vigo, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (5):
  - Jan Sunnegardh's- Private Practice, Gothenburg
  - Universitetssjukhuset i Lund, Lund
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset i Uppsala, Uppsala
  - Universitetssjukhuset i Lund, Uppsala
- United Kingdom (7):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Bristol Royal Hospital for Children, Bristol
  - Medway Maritime Hospital, Gillingham
  - Leeds General Infirmary, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1236 subjects were randomized at 162 sites in 16 countries within the northern hemisphere between 21Oct2005 and 14Dec2005 in Season 1 and 02Oct2007 and 31Dec2007 in Season 2; each subject participated in the study for a single RSV season.
Pre-assignment Details: Subjects were randomized 1:1 on Study Day 0 to receive either 15 mg/kg motavizumab or 15 mg/kg palivizumab. A permuted-block randomization method was used and a separate randomization schedule was generated for each site and cyanotic CHD strata combination.
Groups:
- Motavizumab (MEDI-524): Motavizumab was administered as an intramuscular injection at 15 mg/kg every 30 days during the RSV season for a total of 5 scheduled injections. Additionally, children who underwent cardiac surgery with cardiopulmonary bypass through Study Day 150 were to receive a protocol-specified replacement dose of study drug immediately following the surgery when determined by the physician to be medically stable for an IM injection.
- Palivizumab: Palivizumab was administered as an intramuscular injection at 15 mg/kg every 30 days during the RSV season for a total of 5 scheduled injections. Additionally, children who underwent cardiac surgery with cardiopulmonary bypass through Study Day 150 were to receive a protocol-specified replacement dose of study drug immediately following the surgery when determined by the physician to be medically stable for an IM injection.
Period: Overall Study
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Started | 623 (A subject was randomized without appropriate consent in France and is not included in the results.) | 612
Completed | 604 | 595
Not Completed | 19 | 17
Not completed — Death | 9 | 10
Not completed — Withdrawal of consent | 9 | 7
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motavizumab (MEDI-524) | Palivizumab | Total
Number analyzed (Participants) | 623 | 612 | 1235
Age Continuous [Mean (Standard Deviation); unit: months] | 8.47 (6.40) | 8.18 (6.51) | 8.33 (6.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 298 | 580
  Male | 341 | 314 | 655
Race/Ethnicity, Customized [Number; unit: participants]
  White/Non-hispanic | 540 | 529 | 1069
  Black | 23 | 20 | 43
  Hispanic | 21 | 23 | 44
  Asian | 10 | 8 | 18
  Other | 29 | 32 | 61
Region of Enrollment [Number; unit: participants]
  United States | 155 | 146 | 301
  Spain | 31 | 26 | 57
  Lebanon | 62 | 66 | 128
  Austria | 7 | 7 | 14
  Israel | 67 | 65 | 132
  Russian Federation | 32 | 34 | 66
  United Kingdom | 26 | 31 | 57
  France | 13 | 15 | 28
  Czech Republic | 35 | 39 | 74
  Hungary | 27 | 26 | 53
  Canada | 27 | 22 | 49
  Belgium | 28 | 26 | 54
  Poland | 50 | 49 | 99
  Bulgaria | 18 | 18 | 36
  Germany | 35 | 31 | 66
  Sweden | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events Through Study Day 150
Description: Adverse events were summarized by system organ class (SOC) and preferred term (using MedDRA Version 11.1) overall.
Time Frame: Days 0-150
Population: The Safety population included all subjects who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Number analyzed (Participants) | 618 | 612
participants | 575 | 566

2. Primary Outcome: Number of Subjects Reporting Serious Adverse Events Through Study Day 150
Description: Serious adverse events were those that resulted in death; were life-threatening; resulted in subject hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization and that, based on appropriate medical judgment, may have jeopardized the subject and may have required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Days 0-150
Population: The Safety population included all subjects who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Number analyzed (Participants) | 618 | 612
participants | 292 | 304

3. Primary Outcome: Number of Subjects Reporting Laboratory Adverse Events
Time Frame: Days 0-150
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Number analyzed (Participants) | 618 | 612
participants
  Adrenal insufficiency | 3 | 3
  Alanine aminotranferase increased | 13 | 26
  Anemia | 17 | 14
  Aspartate aminotransferase increased | 3 | 9
  Bacteria sputum indentified | 1 | 1
  Blood alkaline phosphatase increased | 1 | 0
  Blood calcium decreased | 0 | 1
  Blood calcium increased | 2 | 0
  Blood creatinine increased | 0 | 1
  Blood potassium decreased | 1 | 1
  Blood potassium increased | 1 | 1
  Blood sodium abnormal | 0 | 1
  Blood sodium decreased | 1 | 1
  Blood thyroid stimulating hormone increased | 1 | 0
  Blood urea increased | 39 | 34
  Brain natriuretic peptide increased | 1 | 0
  C-reactive protein increased | 0 | 5
  Clostridium difficiline toxin test positive | 1 | 0
  Coagulation test abnormal | 1 | 1
  Haematocrit drecreased | 0 | 1
  Haemaglobin decreased | 0 | 1
  Hepatic enzyme increased | 3 | 3
  Hyperbilirubinemia | 1 | 0
  Hypertransaminasemia | 0 | 1
  Hypothyroidism | 3 | 2
  International normalised ratio decreased | 0 | 1
  International normalised ratio increased | 0 | 2
  Iron deficiency anaemia | 1 | 0
  Liver function test abnormal | 3 | 2
  Mean cell volume decreased | 1 | 0
  Neutropenia | 1 | 0
  Occult blood positive | 1 | 0
  Oxygen saturation decreased | 9 | 4
  Platelet count decreased | 0 | 1
  Renal function test abnormal | 1 | 0
  Thrombocythemia | 1 | 0
  Thrombocytopenia | 1 | 5
  Thyroid function test abnormal | 0 | 1
  Transaminases increased | 0 | 2
  Urine output decreased | 1 | 1
  White blood cell count increased | 1 | 0

4. Secondary Outcome: The Number of Subjects Hospitalized for RSV Infection.
Description: An RSV hospitalization was defined as one of the following: 1) Cardiac/respiratory hospitalization with a positive real-time RT-PCR RSV diagnostic test performed at a central laboratory, or 2) New onset of lower respiratory tract symptoms with an objective measure of worsening respiratory status in an already hospitalized subject with a positive real-time RT-PCR RSV diagnostic test performed at a central laboratory (nosocomial RSV hospitalization), or 3) Death demonstrated to be caused by RSV (based on virologic evidence and either clinical history or autopsy).
Time Frame: Days 0-150
Population: The ITT population is the primary efficacy analysis population and consists of all subjects randomized into the study.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Number analyzed (Participants) | 623 | 612
participants | 12 | 16
Statistical Analysis 1: Comparison: Motavizumab (MEDI-524) vs Palivizumab; Relative risk and confidence interval adjusted for the stratification factor of CHD stratum (cyanotic or other) specified on the CRF; Test type: Superiority or Other; Guess method; Exact conditional binomial method conditioning on the total number of cases with mid-probability adjustment; Risk Ratio (RR) = 0.746, 95% CI 2-sided [0.344 to 1.586]

5. Secondary Outcome: The Number of Subjects With RSV Outpatient MA-LRI for Season 2 Only.
Description: An RSV outpatient MA-LRI was defined as an outpatient medically-attended event designated by the principal investigator as a lower respiratory illness with a positive real-time RT-PCR RSV diagnostic test performed at a central laboratory.
Time Frame: Days 0-150
Population: All subjects who were randomized in Season 2
Measure: Number; unit: participant
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Number analyzed (Participants) | 304 | 310
participant | 3 | 6
Statistical Analysis 1: Comparison: Motavizumab (MEDI-524); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Guess method; Exact conditional binomial method conditioning on the total number of cases with mid-probability adjustment; Risk Ratio (RR) = 0.495, 95% CI 2-sided [0.101 to 1.989]

6. Secondary Outcome: Number of Subjects Who Had Anti-motavizumab Antibodies Detected
Description: ECLA-based method
Time Frame: Days 0-150
Population: Evaluable for ADA Population; includes all motavizumab-treated subjects who received the correct study drug for their first dose and did not receive commercial palivizumab before receiving any study drug.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 605
participants | 9

7. Secondary Outcome: Mean Trough Serum Concentration of Motavizumab at Pre-dose 1
Description: Trough serum concentrations (ug/mL) of motavizumab at pre-dose 1
Time Frame: Pre-dose 1
Population: Evaluable for PK population; all motavizumab-treated subjects who received any study drug and did not received commercial palivizumab. Excludes subjects after cardiopulmonary bypass surgery.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 543
ug/mL | 0.0 (0.0)

8. Secondary Outcome: Mean Trough Serum Concentration of Motavizumab at 30 Days Post-dose 1
Description: Trough serum concentrations (ug/mL) of motavizumab at 30 days post-dose 1
Time Frame: 30 days post-dose 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 521
ug/mL | 46.90 (15.20)

9. Secondary Outcome: Mean Trough Serum Concentration of Motavizumab at 30 Days Post-dose 2
Description: Trough serum concentrations (ug/mL) of motavizumab at 30 days post-dose 2
Time Frame: 30 days post-dose 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 228
ug/mL | 60.94 (25.41)

10. Secondary Outcome: Mean Trough Serum Concentration of Motavizumab at 30 Days Post-dose 3
Description: Trough serum concentrations (ug/mL) of motavizumab at 30 days post-dose 3
Time Frame: 30 days post-dose 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 203
ug/mL | 66.59 (34.51)

11. Secondary Outcome: Mean Trough Serum Concentration of Motavizumab at 30 Days Post-dose 4
Description: Trough serum concentrations (ug/mL) of motavizumab at 30 days post-dose 4
Time Frame: 30 days post-dose 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 203
ug/mL | 77.87 (32.75)

12. Secondary Outcome: Mean Trough Serum Concentrations of Motavizumab in Subjects Who Underwent Cardiac Surgery With Cardiopulmonary Bypass
Description: Subjects who underwent cardiac surgery with cardiopulmonary bypass through Study Day 150 were to have a blood sample taken for determination of study drug concentrations prior to receipt of another dose of study drug immediately following surgery.
Time Frame: Days 0-150
Population: Evaluable for PK following cardiac surgery with cardiopulomonary bypass; all motivizumab treated subjects who underwent cardiac surgery with cardiopulmonary bypass and who received the correct dose regiment.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524)
Number analyzed (Participants) | 127
ug/mL | 48.51 (27.30)

ADVERSE EVENTS:
Time Frame: Day 0 - Day 150
Arm/Group | Motavizumab (MEDI-524) | Palivizumab
Serious Adverse Events (participants affected / at risk) | 292/618 | 304/612
Other Adverse Events (participants affected / at risk) | 553/618 | 540/612
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) (N=618) | Palivizumab (N=612)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1) | 1 (2)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 2 (2)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC ANEURYSM (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 3 (5)
CARDIAC FAILURE (Cardiac disorders) | 5 (7) | 7 (8)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 4 (4) | 5 (6)
CARDIAC PSEUDOANEURYSM (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 2 (2)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 3 (3)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 1 (2)
CYANOSIS (Cardiac disorders) | 9 (9) | 5 (7)
DRESSLER'S SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 1 (1)
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 (3) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2) | 2 (2)
PULMONARY VALVE STENOSIS (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (2)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANOMALOUS PULMONARY VENOUS CONNECTION (Congenital, familial and genetic disorders) | 2 (5) | 2 (2)
AORTIC VALVE ATRESIA (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 5 (5) | 2 (3)
ATRIOVENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 13 (14) | 22 (25)
CHARGE SYNDROME (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CLEFT LIP AND PALATE (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
CLEFT PALATE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
COARCTATION OF THE AORTA (Congenital, familial and genetic disorders) | 3 (4) | 3 (3)
CONGENITAL AORTIC DILATATION (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CONGENITAL CORONARY ARTERY MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
CONGENITAL MITRAL VALVE STENOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CONGENITAL PULMONARY VALVE ATRESIA (Congenital, familial and genetic disorders) | 8 (10) | 14 (17)
CONGENITAL TRICUSPID VALVE ATRESIA (Congenital, familial and genetic disorders) | 8 (11) | 12 (17)
DEVELOPMENTAL GLAUCOMA (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
DOUBLE OUTLET RIGHT VENTRICLE (Congenital, familial and genetic disorders) | 10 (12) | 7 (7)
EBSTEIN'S ANOMALY (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
FALLOT'S TETRALOGY (Congenital, familial and genetic disorders) | 38 (45) | 49 (63)
HEART DISEASE CONGENITAL (Congenital, familial and genetic disorders) | 4 (4) | 9 (10)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HYPOPLASTIC LEFT HEART SYNDROME (Congenital, familial and genetic disorders) | 16 (23) | 18 (22)
HYPOPLASTIC RIGHT HEART SYNDROME (Congenital, familial and genetic disorders) | 2 (3) | 2 (2)
HYPOSPADIAS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
INTERRUPTION OF AORTIC ARCH (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
LEFT VENTRICLE OUTFLOW TRACT OBSTRUCTION (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
MEDIUM-CHAIN ACETYL-COENZYME A DEHYDROGENASE DEFICIENCY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
MITRAL VALVE ATRESIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
MULTIPLE CARDIAC DEFECTS (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
PATENT DUCTUS ARTERIOSUS (Congenital, familial and genetic disorders) | 4 (4) | 2 (2)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
PULMONARY ARTERY ATRESIA (Congenital, familial and genetic disorders) | 4 (4) | 1 (1)
PULMONARY SEQUESTRATION (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
RIGHT VENTRICLE OUTFLOW TRACT OBSTRUCTION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
SCIMITAR SYNDROME (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
SHONE COMPLEX (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
TRANSPOSITION OF THE GREAT VESSELS (Congenital, familial and genetic disorders) | 4 (4) | 6 (6)
TRUNCUS ARTERIOSUS PERSISTENT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
UNIVENTRICULAR HEART (Congenital, familial and genetic disorders) | 9 (10) | 11 (12)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 29 (32) | 36 (38)
DEAFNESS BILATERAL (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
STRABISMUS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (2)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 3 (4)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 (4) | 6 (8)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SPIGELIAN HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (5)
CATHETER RELATED COMPLICATION (General disorders) | 0 (0) | 1 (1)
CYST (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
IRRITABILITY (General disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 5 (6) | 5 (7)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ADENOVIRAL UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ADENOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1) | 2 (2)
BRONCHIOLITIS (Infections and infestations) | 15 (27) | 16 (17)
BRONCHITIS (Infections and infestations) | 12 (16) | 10 (11)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 4 (4) | 6 (6)
CELLULITIS (Infections and infestations) | 0 (0) | 2 (2)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 1 (1)
CROUP INFECTIOUS (Infections and infestations) | 2 (2) | 1 (1)
EAR INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 2 (2) | 0 (0)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ENTEROBACTER BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3)
GASTROENTERITIS (Infections and infestations) | 17 (17) | 18 (19)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 7 (7) | 14 (14)
GASTROENTERITIS VIRAL (Infections and infestations) | 5 (5) | 6 (6)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 2 (2)
LOBAR PNEUMONIA (Infections and infestations) | 3 (3) | 1 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 4 (4)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1)
LYMPHANGITIS (Infections and infestations) | 0 (0) | 1 (1)
MEDIASTINITIS (Infections and infestations) | 1 (1) | 2 (2)
MENINGITIS MENINGOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (3) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 5 (5) | 1 (1)
OTITIS MEDIA ACUTE (Infections and infestations) | 2 (2) | 1 (1)
OTITIS MEDIA VIRAL (Infections and infestations) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 3 (3)
PHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA (Infections and infestations) | 20 (27) | 23 (24)
PNEUMONIA ADENOVIRAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 6 (6) | 9 (9)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 2 (2) | 4 (4)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 4 (4)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 (2) | 1 (1)
RHINITIS (Infections and infestations) | 1 (1) | 0 (0)
ROTAVIRUS INFECTION (Infections and infestations) | 1 (1) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL MEDIASTINITIS (Infections and infestations) | 1 (1) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TRACHEITIS (Infections and infestations) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (12) | 11 (12)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 2 (2)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 1 (1) | 1 (1)
VARICELLA (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 1 (1)
VIRAL SINUSITIS (Infections and infestations) | 1 (2) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
AORTIC INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SHUNT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SHUNT STENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1)
CENTRAL VENOUS PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0)
COAGULATION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 2 (2)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
MEDICAL OBSERVATION (Investigations) | 2 (2) | 1 (2)
SLEEP STUDY (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
DIET REFUSAL (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
FEEDING DISORDER (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FEEDING DISORDER OF INFANCY OR EARLY CHILDHOOD (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
WEIGHT GAIN POOR (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
SOFT TISSUE NECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 2 (2) | 1 (1)
FEBRILE CONVULSION (Nervous system disorders) | 1 (1) | 1 (1)
MYOCLONUS (Nervous system disorders) | 0 (0) | 1 (1)
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
TONIC CLONIC MOVEMENTS (Nervous system disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
PYELOCALIECTASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
APNOEIC ATTACK (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOPULMONARY DYSPLASIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DIAPHRAGM MUSCLE WEAKNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DIAPHRAGMATIC HERNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
LARYNGEAL GRANULOMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY ARTERY STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
PULMONARY HYPERTENSIVE CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
PULMONARY VEIN OCCLUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY VEIN STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TRACHEOMALACIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SOCIAL STAY HOSPITALISATION (Social circumstances) | 2 (2) | 0 (0)
IMMUNISATION (Surgical and medical procedures) | 1 (1) | 0 (0)
URETHRAL MEATOTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 3 (3) | 1 (1)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
VASOSPASM (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) (N=618) | Palivizumab (N=612)
ANAEMIA (Blood and lymphatic system disorders) | 14 (15) | 16 (22)
CARDIAC FAILURE (Cardiac disorders) | 9 (10) | 10 (10)
CYANOSIS (Cardiac disorders) | 25 (42) | 25 (32)
CONJUNCTIVITIS (Eye disorders) | 39 (42) | 27 (32)
CONSTIPATION (Gastrointestinal disorders) | 44 (47) | 31 (35)
DIARRHOEA (Gastrointestinal disorders) | 69 (80) | 64 (70)
FLATULENCE (Gastrointestinal disorders) | 5 (5) | 6 (7)
ENTERITIS (Gastrointestinal disorders) | 7 (8) | 4 (4)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 19 (19) | 23 (23)
TEETHING (Gastrointestinal disorders) | 44 (54) | 36 (56)
VOMITING (Gastrointestinal disorders) | 59 (70) | 49 (60)
IRRITABILITY (General disorders) | 22 (33) | 37 (48)
PYREXIA (General disorders) | 180 (285) | 177 (286)
IMMUNISATION REACTION (Immune system disorders) | 6 (8) | 8 (11)
BRONCHIOLITIS (Infections and infestations) | 16 (18) | 10 (11)
BRONCHITIS (Infections and infestations) | 40 (48) | 41 (57)
CANDIDIASIS (Infections and infestations) | 6 (6) | 5 (7)
CROUP INFECTIOUS (Infections and infestations) | 2 (2) | 9 (9)
EAR INFECTION (Infections and infestations) | 9 (11) | 7 (9)
EXANTHEMA SUBITUM (Infections and infestations) | 6 (6) | 7 (7)
GASTROENTERITIS (Infections and infestations) | 56 (62) | 48 (53)
GASTROENTERITIS VIRAL (Infections and infestations) | 9 (9) | 5 (5)
INFLUENZA (Infections and infestations) | 6 (6) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (12) | 9 (13)
NASOPHARYNGITIS (Infections and infestations) | 67 (83) | 57 (79)
ORAL CANDIDIASIS (Infections and infestations) | 10 (10) | 7 (11)
OTITIS MEDIA (Infections and infestations) | 73 (97) | 70 (95)
OTITIS MEDIA ACUTE (Infections and infestations) | 26 (30) | 19 (25)
PHARYNGITIS (Infections and infestations) | 31 (37) | 24 (28)
PNEUMONIA (Infections and infestations) | 11 (12) | 13 (14)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (12) | 4 (5)
RHINITIS (Infections and infestations) | 91 (115) | 77 (99)
SINUSITIS (Infections and infestations) | 10 (11) | 7 (8)
TONSILLITIS (Infections and infestations) | 18 (21) | 8 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 160 (235) | 164 (254)
URINARY TRACT INFECTION (Infections and infestations) | 12 (13) | 9 (9)
VARICELLA (Infections and infestations) | 11 (11) | 5 (5)
VIRAL INFECTION (Infections and infestations) | 38 (47) | 30 (33)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (13) | 15 (16)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 13 (13) | 25 (25)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 9 (9)
BLOOD UREA INCREASED (Investigations) | 39 (39) | 34 (35)
OXYGEN SATURATION DECREASED (Investigations) | 9 (10) | 4 (5)
WEIGHT DECREASED (Investigations) | 7 (7) | 6 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (5) | 6 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 (6) | 5 (6)
RESTLESSNESS (Psychiatric disorders) | 6 (7) | 3 (3)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 92 (120) | 71 (95)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 33 (45)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (7)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 28 (35)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 49 (64) | 45 (70)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (12)
DERMATITIS (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 32 (38) | 31 (38)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 11 (13) | 9 (9)
RASH (Skin and subcutaneous tissue disorders) | 27 (27) | 21 (25)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 9 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.